CLINICAL TRIAL: NCT04181515
Title: Using Repetitive Transcranial Magnetic Stimulation (rTMS) to Explore Neural Mechanisms of Stress-Induced Opioid Use
Brief Title: Using rTMS to Explore Neural Mechanisms of Stress-Induced Opioid Use
Acronym: OTC-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OTC-1
Record Dates: First submitted 2019-11-24; First posted 2019-11-29 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Stress; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Yohimbine; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: mixed design, with 4 (2x2) within-subject conditions (placebo vs. stressor X sham vs. rTMS), each occurring in two parallel groups (10 Hz dorsolateral prefrontal cortex vs. sham rTMS in group 1, and 1 Hz medial prefrontal cortex vs. sham rTMS in group 2)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: placebo for stressor, and sham figure of 8 coil for rTMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- placebo stressor, sham rTMS (Placebo Comparator): placebo stressor (lactose), sham rTMS (inactive coil)
  Interventions: Drug: Placebo oral tablet; Device: sham rTMS
- placebo stressor, active rTMS (Active Comparator): placebo stressor (lactose), active rTMS (10 Hz dlPFC in group 1; 1 Hz mPFC in group 2)
  Interventions: Drug: Placebo oral tablet; Device: active rTMS
- stressor, sham rTMS (Active Comparator): stressor (yohimbine 54mg + hydrocortisone 20mg), sham rTMS (inactive coil)
  Interventions: Drug: Yohimbine + Hydrocortisone; Device: sham rTMS
- stressor, active rTMS (Active Comparator): stressor (yohimbine 54mg + hydrocortisone 20mg), active rTMS (10 Hz dlPFC in group 1; 1 Hz mPFC in group 2)
  Interventions: Drug: Yohimbine + Hydrocortisone; Device: active rTMS

INTERVENTIONS:
Drug: Placebo oral tablet — placebo stressor
  Arms: placebo stressor, active rTMS; placebo stressor, sham rTMS
Drug: Yohimbine + Hydrocortisone — Yohimbine 54mg + Hydrocortisone 20mg
  Arms: stressor, active rTMS; stressor, sham rTMS
Device: sham rTMS — sham rTMS (inactive coil)
  Arms: placebo stressor, sham rTMS; stressor, sham rTMS
Device: active rTMS — active rTMS (10 Hz dlPFC stimulation in group 1; 1 Hz mPFC stimulation in group 2)
  Arms: placebo stressor, active rTMS; stressor, active rTMS

SUMMARY:
This study will use a stress (vs. placebo) exposure model, paired with single-session sham vs. active rTMS at two distinct cortical locations (dlPFC vs. mPFC in parallel groups) to assess whether rTMS neuromodulation at these alternative loci differentially influence stress-reactivity and opioid reinforcement in non-treatment seeking participants with OUD. Stress-reactivity will be measured using cognitive, affective, behavioral and biological phenotypes.

DETAILED DESCRIPTION:
The Competing Neurobehavioral Decisions Systems (CNDS) model of addiction suggests that persons with SUDs have hyperactive limbic reward circuitry and hypoactive executive control circuitry. CNDS theory supports targeting the dorsolateral prefrontal cortex (dlPFC, part of executive control circuit) and other cortical targets with repetitive transcranial magnetic stimulation (rTMS). One candidate-the medial prefrontal cortex (mPFC)-is part of limbic reward circuitry and accessible using rTMS. We validated a rigorous pharmacological stress-induction method (yohimbine + hydrocortisone) that emulates endogenous stress-reactivity and have established linkages between stress-exposure, executive dysfunction, and drug seeking. Our lab is developing rTMS as a potential "anti-stress" neuromodulation approach in people with opioid use disorder (OUD).

This study will use a stress (vs. placebo) exposure model, paired with single-session sham vs. active rTMS at two distinct cortical locations (dlPFC vs. mPFC in parallel groups) to assess whether rTMS neuromodulation at these alternative cortical loci differentially influence stress-reactivity and opioid reinforcement in non-treatment seeking participants with OUD. Stress-reactivity will be measured using cognitive, affective, behavioral and biological phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for OUD
* Age 21-60 yr
* Right handed
* Males and non-pregnant/non-lactating females
* Cognitively intact (total IQ score >80 on Shipley Institute of Living Scale
* Screening cardiovascular indices within ranges for safe use of the pharmacological stressor: resting HR 50-90 bpm, systolic BP 90-140 mmHg, and diastolic BP 50-90 mmHg
* Use alcohol and/or marijuana <3 times/week; each "time" should consist of <1 marijuana "joint" equivalent and <3 alcoholic drinks.

Exclusion Criteria:

* Under influence of any substance during session
* Past 7-day use of illicit drugs other than opioids (except marijuana, which is legal in Michigan)
* Urinalysis positive for cocaine metabolites, benzodiazepines, barbiturates, amphetamines or pregnancy
* Medical conditions prohibiting use of rTMS (e.g. seizure history; based on rTMS screening questionnaire)
* Lifetime diagnosis of: psychotic disorder, bipolar disorder, generalized anxiety disorder, or obsessive compulsive disorder; major depression in the past 5 years; or potentially antisocial personality disorder (if the clinical psychologist judges such behaviors to be potentially disruptive or unsafe in our lab)
* Past-year SUD other than OUD
* Acute/unstable illness: conditions making it unsafe for participation (e.g. neurological, cardiovascular, pulmonary, or systemic diseases)
* Lactose intolerance (placebo dose)
* Any prohibited medications: medications that lower seizure threshold, psychiatric medications, prescription pain medications, or blood pressure medications
* Chronic head or neck pain
* Past-month participation in a research study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Addiction Stroop task | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  reaction time (msec) measure of cognitive interference
Digit Span Task | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  number of digits recalled, measure of verbal working memory
Wisconsin Card Sorting Task | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  number of correct items, measures ability to shift set and assesses cognitive flexibility
Monetary Incentive Delay task | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  number of rewards received, measure of motivation
Delay Discounting task | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  rate of monetary discounting
Drug/Money Choice Task | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  number of hypothetical choices between a constant amount of preferred opioid (relative to money)
Blood pressure | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Systolic/diastolic BP (mm Hg)
Heart rate | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Heart rate (beats/min)
Saliva cortisol level | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Saliva cortisol level (µg/dL)
Saliva alpha-amylase level | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Saliva alpha-amylase level (U/mL)
Serum prolactin level | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Serum prolactin level (pg/dL)
Serum BDNF level | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Serum brain derived neurotrophic factor level (pg/dL)
Positive and Negative Affect Schedule (PANAS) positive affect | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  10-item sub scale score of positive affect
Positive and Negative Affect Schedule (PANAS) negative affect | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  10-item sub scale score of negative affect
State Trait Anxiety Inventory | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  state anxiety scores
Desire for Drug Questionnaire | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  opioid craving score
Opiate-32 Questionnaire, Agonist score | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  total opioid agonist score (16 items)
Opiate-32 Questionnaire, Withdrawal score | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  total opioid withdrawal symptom score (16 items)
Resting-state EEG activation | change from pre- and post-intervention in each of 4 sessions (through study completion, about 1 month total)
  relative (gamma band ÷ slow band) ratio in electroencephalogram (EEG) power during resting state

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, qualified investigators may apply in writing to receive the study protocol. At this time, it has not been determined whether data will be shared and the conditions for access.
Supporting Information: Study Protocol
Time Frame: Available after the study is completed
Access Criteria: Qualified investigators may apply in writing.